CLINICAL TRIAL: NCT07320729
Title: Can Intraoral Photogrammetry Overcome Surgical Field Challenges? An In-Vivo Accuracy Study in Immediate Full-Arch Loading
Brief Title: Accuracy of Intraoral Photogrammetry vs Optical Scanners for Immediate Full-Arch Implant Loading
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abdelrahman Khalaf Eldabe (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Khalaf Eldabe, Lecturer of Oral Medicine and Periodontology , Assiut University, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-2025-00027
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Edentulism; Implant-supported Full-arch Prosthesis; Digital Impression Accuracy; Photogrammetry in Dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraoral Optical Scanner (IOS) (Experimental): Participants will undergo a digital implant impression using a conventional intraoral optical scanner immediately after implant placement to capture implant positions for immediate full-arch loading.
  Interventions: Device: Intraoral Optical Scanner
- Intraoral Photogrammetry Scanner (IPS) (Experimental): Participants will undergo a digital implant impression using an intraoral photogrammetry scanner immediately after implant placement to capture implant coordinates using photogrammetric scan flags combined with intraoral soft tissue scanning.
  Interventions: Device: Intraoral Photogrammetry Scanner Elite (Shining3D)

INTERVENTIONS:
Device: Intraoral Optical Scanner — Digital intraoral scanning of implant positions using standard scan bodies for complete-arch implant impressions.
  Arms: Intraoral Optical Scanner (IOS)
Device: Intraoral Photogrammetry Scanner Elite (Shining3D) — Intraoral photogrammetric capture of implant coordinates using scan flags, combined with soft tissue scanning, without stitching.
  Arms: Intraoral Photogrammetry Scanner (IPS)

SUMMARY:
This prospective in vivo clinical trial evaluates and compares the accuracy (trueness) and scanning time of intraoral photogrammetry scanners (IPS) versus conventional intraoral optical scanners (IOS) for immediate full-arch implant impressions. The reference standard will be a verified conventional splinted open-tray impression taken at the uncovering stage. Sixty edentulous arches receiving 4-6 implants will be included. Linear, angular, and 3D Euclidean deviations will be calculated to assess accuracy.

DETAILED DESCRIPTION:
Digital impression systems are widely used for implant dentistry, but complete-arch implant scans remain challenging due to lack of stable landmarks and intraoral movement. Photogrammetry technology captures implant coordinates with high trueness by eliminating stitching errors and excluding unstable soft tissue. A newly introduced intraoral photogrammetry scanner (IPS) integrates photogrammetry and intraoral imaging in a single device.

This study is the first in-vivo prospective clinical trial comparing IOS and IPS accuracy in immediate complete-arch implant loading. Patients receiving 4-6 implants in one arch will undergo two digital impressions immediately after surgery: one using IOS (AoralScan 3) and one using IPS (Elite). A conventional splinted open-tray impression at second-stage surgery will be used as the reference model. Digital files will be superimposed to calculate linear, angular, and 3D (Euclidean) deviations. Scanning time and effect of arch type will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Completely edentulous arch to receive 4-6 implants. Candidate for immediate loading with a one-piece fixed prosthesis. ASA I or II medically healthy patients. Patient able to attend follow-up visits and sign informed consent.

Exclusion Criteria:

Medically compromised patients (ASA III or higher). Poor oral hygiene or heavy smokers. Insufficient bone volume for implant placement. Uncooperative patients or those refusing participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-12-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Trueness of Implant Position (3D Euclidean Deviation) | 3 Months
  The primary outcome is to evaluate the clinical performance of conventional intraoral scanners (IOS) and intraoral photogrammetry scanners (IPS) in immediate complete arch implant loading for each patient enrolled in the study, with a paired comparison of the deviation differences (Degree of Trueness).

SECONDARY OUTCOMES:
Effect of Arch Type on Digital Impression Trueness | 3 Months
  The secondary outcome is to analyze the potential effect (correlation) of the type of arch (maxilla vs. mandible) on the degree of trueness. Also, the scanning time of the 2 techniques will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt